CLINICAL TRIAL: NCT07007494
Title: The Relationship Between Preoperative Nutritional and Inflammatory Markers and Early Postoperative Clinical Outcomes in Patients Undergoing Bariatric Surgery
Brief Title: Early Outcomes and Nutritional Scores in Bariatric Patients
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Istinye University
Other Study IDs: PNI HALP OBESITY
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Complications; Preoperative Nutritional Markers
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nutritional and Inflammatory Marker Evaluation — This is a prospective observational cohort study evaluating whether preoperative immune-nutritional markers-including Prognostic Nutritional Index (PNI), HALP score, Neutrophil-to-Lymphocyte Ratio (NLR), and C-Reactive Protein (CRP)-can predict early postoperative clinical outcomes (complication development, time to oral intake, mobilization, and length of hospital stay) in patients undergoing elective laparoscopic sleeve gastrectomy. No intervention or treatment is administered as part of this study. All data are collected from routine preoperative laboratory tests and standard postoperative clinical follow-up.

SUMMARY:
This prospective observational study aims to evaluate whether preoperative immune-nutritional markers-specifically the Prognostic Nutritional Index (PNI), HALP score, Neutrophil-to-Lymphocyte Ratio (NLR), and C-Reactive Protein (CRP)-can predict early postoperative clinical outcomes such as time to oral intake, mobilization, complications, and length of hospital stay in patients undergoing elective laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Body mass index (BMI) ≥ 35 kg/m²
* Scheduled for elective laparoscopic sleeve gastrectomy
* Availability of complete preoperative laboratory test results
* Signed informed consent

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Presence of active infection
* History of immunosuppressive therapy or hematologic malignancy
* Need for intensive care unit (ICU) admission within the first 72 hours postoperatively
* Preoperative administration of albumin or blood products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years with morbid obesity (BMI ≥ 35 kg/m²) who are scheduled to undergo elective laparoscopic sleeve gastrectomy at a tertiary care center.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Postoperative Complications Within 72 Hours | Up to 72 hours after surgery
  Complications such as fever, surgical site infection, nausea/vomiting, hypotension, or need for reintervention will be recorded during the first 72 hours after laparoscopic sleeve gastrectomy. The association between preoperative nutritional and inflammatory scores (PNI, HALP, NLR, CRP) and complication occurrence will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Courcoulas AP, Daigle CR, Arterburn DE. Long term outcomes of metabolic/bariatric surgery in adults. BMJ. 2023 Dec 18;383:e071027. doi: 10.1136/bmj-2022-071027. PMID 38110235
- [Result] Ishiguro T, Aoyama T, Ju M, Kazama K, Fukuda M, Kanai H, Sawazaki S, Tamagawa H, Tamagawa A, Cho H, Hara K, Numata M, Hashimoto I, Maezawa Y, Segami K, Oshima T, Saito A, Yukawa N, Rino Y. Prognostic Nutritional Index as a Predictor of Prognosis in Postoperative Patients With Gastric Cancer. In Vivo. 2023 May-Jun;37(3):1290-1296. doi: 10.21873/invivo.13207. PMID 37103068
- [Result] Xu F, Meng C, Yang Z, Li H, Gao J, Sun L, Zhang X, Wei Q, Wu G, Yao H, Zhang Z. Prognostic nutrition index predicts short-term surgical complications in patients with rectal cancer after laparoscopic surgery. Front Surg. 2022 Oct 25;9:1000108. doi: 10.3389/fsurg.2022.1000108. eCollection 2022. PMID 36386497
- [Result] Lee JY, Kim HI, Kim YN, Hong JH, Alshomimi S, An JY, Cheong JH, Hyung WJ, Noh SH, Kim CB. Clinical Significance of the Prognostic Nutritional Index for Predicting Short- and Long-Term Surgical Outcomes After Gastrectomy: A Retrospective Analysis of 7781 Gastric Cancer Patients. Medicine (Baltimore). 2016 May;95(18):e3539. doi: 10.1097/MD.0000000000003539. PMID 27149460
- [Result] Demirpolat MT, Sisik A. Effectiveness of the Modified Hemoglobin, Albumin, Lymphocyte, and Platelet Score in Predicting Weight Loss After Laparoscopic Sleeve Gastrectomy. J Laparoendosc Adv Surg Tech A. 2024 Jan;34(1):61-66. doi: 10.1089/lap.2023.0333. Epub 2023 Oct 25. PMID 37878772
- [Result] Radkhah H, Zooravar D, Shateri-Amiri B, Saffar H, Najjari K, Hazaveh MM. Predictive Value of Complete Blood Count (CBC)-Derived Indices-C-Reactive-Protein-Albumin-Lymphocyte index (CALLY), Glucose-to-Lymphocyte Ratio (GLR), Prognostic Nutritional Index (PNI), Hemoglobin, Albumin, Lymphocyte, Platelet (HALP), and Controlling Nutritional Status (COUNT)-on Body Composition Changes After Bariatric Surgery. Obes Surg. 2025 Feb;35(2):544-555. doi: 10.1007/s11695-024-07643-1. Epub 2025 Jan 8. PMID 39775392